CLINICAL TRIAL: NCT02138435
Title: Cardiac Output During Exercise in Young Adults Operated for Ventricular Septal Defect as Children
Brief Title: Longterm Outcome After Ventricular Septal Defect Closure
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: VSDBAA2014; 2007-58-0010 (Other: The Danish Data Protection Agency); 1-10-72-7-14 (Other: The Regional Committee on Biomedical Research Ethics)
Record Dates: First submitted 2014-05-01; First posted 2014-05-14 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-09

CONDITIONS: Ventricular Septal Defect
MeSH Terms: conditions — Heart Septal Defects, Ventricular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- VSD-patients: Patients who had VSD closure between 1990 and 1995. They will be tested by a MRI exercise test and a gas-exchange exercise test measuring cardiac output.
  Interventions: Other: MRI exercise test; Other: Gas-exchange exercise test
- Control: A group of healthy control subjects. They will be tested by a MRI exercise test and a gas-exchange exercise test measuring cardiac output.
  Interventions: Other: MRI exercise test; Other: Gas-exchange exercise test

INTERVENTIONS:
Other: MRI exercise test — Measuring cardiac output with MRI during exercise on an ergometer bicycle.
Other: Gas-exchange exercise test — Measuring cardiac output by gas-exchange, while during exercise on an ergometer bicycle.

SUMMARY:
Isolated ventricular septal defect (VSD) is a well know congenital heart anomaly. If discovered in infancy or early childhood surgical intervention can be of necessity depending on the size of the defect, to assure a healthy adulthood. The long-term results of surgical closure of VSD in childhood are good and after surgery the children are considered as equally healthy and physically fit as their peers. However, there is inconsistency in data regarding follow-up on this group of patients, in relation to exercise capacity as a measure of the cardiopulmonary function. To further approach this matter the post-operative cardiac factors of these patients have to be investigated.

With this study the investigators intend to examine the long-term outcome on cardiac output after heart surgery in VSD-patients. It presents an opportunity to also evaluate the correlation between cardiac output determined by gas-exchange and by MRI. The overall objectives of this study are to 1) examine whether VSD-operated patients have reduced cardiac output during exercise in comparison with matched controls, and furthermore 2) to evaluate a correlation between cardiac output measured by MRI and cardiac output determined by gas-exchange.

The project is designed as a long-term follow-up and method study. A cohort of 20 children who in the 1990's underwent surgical closure of a congenital VSD will be asked to participate in this study. An equal amount of healthy young adults, will function as control group. Each participant will complete two different exercise tests, a MRI of the heart during lower body exercise on a supine ergometer bicycle, and a Supine ergometer bicycle exercise test. This data can be used for comparing cardiac output between the test groups, and furthermore it allows an evaluation of the correlation between the two methods.

VSD is as described, the most common congenital heart anomaly. If not intervened with in childhood, it can cause severe heart complications later in life. It is unclear whether this intervention can cause long-term impact on patients exercise capacity, and for that reason it is of great importance that we strive for improving our knowledge of the long-term postsurgical outcome after VSD-closure.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Surgical correction of VSD between 1990 and 1995
* Controls: 18-25 years old, with no medical records of heart disease

Exclusion Criteria:

* Missing journal
* Operation by ventriculotomy
* Other congenital anomalies
* Metallic implants or foreign objects
* Pregnancy

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Of 182 children who in the years 1990 to 1995 underwent surgical closure of a congenital VSD at Aarhus University Hospital (AUH), Denmark, a small group of 20 is randomly selected to participate. These children form a homogenous group of patients comparing surgeons, anesthetists, surgical procedures and post-surgical period. An equal amount of healthy controls, matched on age and gender, form the control group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Cardiac Output | 20 years after VSD surgery
  MRI measured: From obtained standard scout images of the heart and great vessels, flow measurement planes will be planned orthogonally to the ascending aorta and the pulmonary artery. MRI real-time flow will then be measured at different exercise levels orthogonally to the ascending aorta and pulmonary artery just above the level of the valves. Ascending aortic and pulmonary artery blood flow will be used to measure cardiac output in post-MRI analysis.
  Gas-exchange measured: Using a supine ergometer cycle, the pulmonary ventilation and gas exchange will be measured breath-by-breath. End points are peak oxygen uptake, stroke volume, and cardiac output. Fick's principle will be used for estimating cardiac output.

SECONDARY OUTCOMES:
Correlation | 20 years after VSD surgery
  Correlation between MRI measured cardiac output and gas-exchange measured cardiac output.

CONTACTS AND LOCATIONS:
Overall Officials: Vibeke E Hjortdal, Prof., DMSc, Principal Investigator — Aarhus University Hospital
Locations (1):
- Department of Cardiothoracic surgery, Aarhus University Hospital, Aarhus, Denmark

REFERENCES:
- [Background] Heiberg J, Laustsen S, Petersen AK, Hjortdal VE. Reduced long-term exercise capacity in young adults operated for ventricular septal defect. Cardiol Young. 2015 Feb;25(2):281-7. doi: 10.1017/S1047951113002084. Epub 2013 Nov 21. PMID 24565413
- [Background] Meijboom F, Szatmari A, Utens E, Deckers JW, Roelandt JR, Bos E, Hess J. Long-term follow-up after surgical closure of ventricular septal defect in infancy and childhood. J Am Coll Cardiol. 1994 Nov 1;24(5):1358-64. doi: 10.1016/0735-1097(94)90120-1. PMID 7930261
- [Background] Binkhorst M, van de Belt T, de Hoog M, van Dijk A, Schokking M, Hopman M. Exercise capacity and participation of children with a ventricular septal defect. Am J Cardiol. 2008 Oct 15;102(8):1079-84. doi: 10.1016/j.amjcard.2008.05.063. Epub 2008 Jul 26. PMID 18929713
- [Background] Reybrouck T, Rogers R, Weymans M, Dumoulin M, Vanhove M, Daenen W, Van der Hauwaert L, Gewillig M. Serial cardiorespiratory exercise testing in patients with congenital heart disease. Eur J Pediatr. 1995 Oct;154(10):801-6. doi: 10.1007/BF01959785. PMID 8529676
- [Background] Pedersen LM, Pedersen TA, Pedersen EM, Hojmyr H, Emmertsen K, Hjortdal VE. Blood flow measured by magnetic resonance imaging at rest and exercise after surgical bypass of aortic arch obstruction. Eur J Cardiothorac Surg. 2010 Mar;37(3):658-61. doi: 10.1016/j.ejcts.2009.07.041. Epub 2009 Sep 16. PMID 19762252
- [Background] Hjortdal VE, Christensen TD, Larsen SH, Emmertsen K, Pedersen EM. Caval blood flow during supine exercise in normal and Fontan patients. Ann Thorac Surg. 2008 Feb;85(2):599-603. doi: 10.1016/j.athoracsur.2007.08.062. PMID 18222273